CLINICAL TRIAL: NCT07081633
Title: An Open-label, Multi-center Phase II Study of Durvalumab and Tremelimumab With Lenvatinib as First-line Treatment in Patients With Unresectable Hepatocellular Carcinoma
Brief Title: Durvalumab and Tremelimumab With Lenvatinib as First-line Treatment in Patients With Unresectable Hepatocellular Carcinoma
Acronym: TREMENDOUS-2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D419CL00025
Record Dates: First submitted 2025-06-23; First posted 2025-07-23 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — durvalumab; tremelimumab; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): Durvalumab and Tremelimumab with Lenvatinib
  Interventions: Drug: Durvalumab; Drug: Tremelimumab; Combination Product: Lenvatinib

INTERVENTIONS:
Drug: Durvalumab — Durvalumab IV (intravenous infusion)
  Other Names: MEDI4736
Drug: Tremelimumab — Tremelimumab IV (intravenous infusion)
Combination Product: Lenvatinib — Lenvatinib Oral

SUMMARY:
This is a Phase II, single-arm, multicentre study, assessing the efficacy and safety of durvalumab and tremelimumab with lenvatinib in participants with unresectable HCC.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HCC based on histopathological findings from tumor tissues or radiologically findings.
* Must not have received prior systemic therapy for unresectable HCC.
* Barcelona Clinic Liver Cancer (BCLC) stage B (that is not eligible for locoregional therapy) or stage C.
* Child-Pugh Score class A.
* ECOG performance status of 0 or 1 at enrollment.
* At least 1 measurable lesion per RECSIT 1.1 guidelines

Exclusion Criteria:

* Any unresolved toxicity National Cancer Institute (NCI) Common Terminology Criteria for Adverse Event (CTCAE) Grade ≥2 from previous anticancer therapy.
* History of hepatic encephalopathy within past 12 months or requirement for medications to prevent or control encephalopathy.
* Clinically meaningful ascites.
* Patients with main portal vein thrombosis.
* Active or prior documented GI bleeding.
* Patient currently exhibits symptomatic or uncontrolled hypertension.
* Patients co-infected with HBV and HCV, or co-infected with HBV and hepatitis D virus (HDV)
* Uncontrolled intercurrent illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) per RECIST 1.1 | From the date of first dose until the date of objective PD per RECIST 1.1 or death, whichever came first. It will be assessed when approximately 69 PFS events have occurred (60% maturity), approximately 8 months after the last patients dosed.
  Efficacy endpoint

SECONDARY OUTCOMES:
Grade ≥ 3 TRAE within 6 months after the initiation of study intervention | From first dose to 6 months after the initiation of study intervention
  safety endpoint
Overall Survival (OS) | From the date of the first dose of study intervention until death due to any cause. It will be assessed when approximately 69 OS events have occurred (60% maturity), approximately 24 months after last participant has been assigned to study intervention.
  Efficacy endpoint
Objective Response Rate (ORR) per RECIST 1.1 | From the date of the first dose of study intervention until the date of objective PD per RECIST 1.1. It is anticipated that this analysis will be performed approximately 8 months after the last patient has been assigned to study intervention.
  Efficacy endpoint
Disease Control Rate (DCR) per RECIST 1.1 | From the date of the first dose of study intervention until the date of objective PD per RECIST 1.1. It is anticipated that this analysis will be performed approximately 8 months after the last patient has been assigned to study intervention.
  Efficacy endpoint
Duration of response (DoR) per RECIST 1.1 | From the date of response until the date of objective PD per RECIST 1.1 or death, whichever came first. It is anticipated that this analysis will be performed approximately 8 months after the last patient dosed.
  Efficacy endpoint
Progression Free Survival (PFS) per mRECIST | From the date of the first dose until the date of objective PD per mRECIST or death, whichever came first. It will be assessed when approximately 69 PFS events have occurred (60% maturity), approximately 8 months after the last patients dosed.
  Efficacy endpoint

CONTACTS AND LOCATIONS:
Locations (17):
- China (16):
  - Research Site, Beijing
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Jinan
  - Research Site, Nanjing
  - Research Site, Ningbo
  - Research Site, Shanghai
  - Research Site, Taiyuan
  - Research Site, Tianjin
  - Research Site, Wenzhou
  - Research Site, Wuhan
  - Research Site, Xiamen
  - Research Site, Zhengzhou
- Research Site, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient- level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  Plan Description: All request will be evaluated as per the Az disclosure commitment:
  https://astrazenecaarouptrials.pharmacm.com/ST/Submission/Disclosure Yes. indicates that Az are accepting requests for IPD ,but this does not mean are quests will be shared
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitment at made to the EFPIA Pharma Data Sharing Principles .For details of our timeline please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool.
  Signed Data Sharing Agreement(non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to a air access. For additional details. please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home